CLINICAL TRIAL: NCT04983355
Title: Efficacy of the Marine Based Nutritional Supplement Peptidyss® on Sleep and Anxiety : a Randomized Clinical Trial With a Cross-Over Design in Healthy Adults
Brief Title: Efficacy of the Marine Based Nutritional Supplement Peptidyss® on Sleep and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abyss Ingredients (Industry)
Collaborators: Daacro (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PEPTIDYSS
Record Dates: First submitted 2021-07-07; First posted 2021-07-30 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Sleep Disorder
Keywords: sleep disorder; anxiety; stress; fish hydrolysate; food supplement
MeSH Terms: conditions — Sleep Wake Disorders; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peptidyss (Experimental): Dietary supplement : fish hydrolysate
  The experimental product is a dietary supplement composed of a hydrolysate of fish containing low molecular weight peptides (4 capsules/day providing 1,4 g of fish hydrolysate)
  Interventions: Dietary Supplement: Fish Hydrolysate
- Placebo (Placebo Comparator): The placebo product containing mainly silica is presented in the same form as the active product, so that people handling the product cannot distinguish both formula (4 capsules/day)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fish Hydrolysate — The participants take 4 capsules/day of the study product. Two capsules should be consumed orally every morning with breakfast and/or with a glass of (plain, not sparkling) water and not with fruit juice or hot food/drink while ingesting the capsules; and two capsules should be consumed orally every evening with their dinner and/or with a glass of water.
  Participants receiving the fish hydrolysate the fourth first weeks will then receive the placebo during another 4 weeks. A wash-out period of 4 weeks is included between each phase of supplementation.
  Arms: Peptidyss
Dietary Supplement: Placebo — The participants take 4 capsules/day of the study product. Two capsules should be consumed orally every morning with breakfast and/or with a glass of (plain, not sparkling) water and not with fruit juice or hot food/drink while ingesting the capsules; and two capsules should be consumed orally every evening with their dinner and/or with a glass of water.
  Participants receiving the Placebo the fourth first weeks will then receive the fish hydrolysate during another 4 weeks. A wash-out period of 4 weeks is included between each phase of supplementation.
  Arms: Placebo

SUMMARY:
This interventional, double-blind, randomized, placebo-controlled pilot study aims to evaluate the effect of a dietary supplementation of a fish hydrolysate Peptidyss on sleep quality and anxiety.

DETAILED DESCRIPTION:
A total of 44 healthy participants (n=22 female, n=22 male) aged 35-60 years inclusive are included into the study, in a cross-over design. The participants will take both products, the fish hydrolysate Peptidyss and the placebo during a period of 4 weeks per product. The total duration of the study per participant is 127 days. The study visits are defined as Screening Visit and Study Inclusion (V0), Pre-Intervention-1-Visit (V1), Post-Intervention-1-Visit (V2), Follow-up-Intervention-1-Visit / Pre-Intervention-2-Visit (V3), Post-Intervention-2-Visit (V4) and Follow-up-Intervention-2-Visit (V5). The 4 weeks between V2 and V3 will serve as a washout phase between Intervention-1 and Intervention-2. No further follow-up visit is planned.

The primary objective is to evaluate the efficacy of Peptidyss® on sleep quality.

The secondary objectives are to evaluate the efficacy of Peptidyss® on sleep quality, anxiety, perceived stress and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary, written, informed consent to participate in the study
* Male or female aged between 35-60 years (inclusive)
* Body mass index (BMI) between ≥18.0 - ≤35.0 kg/m2
* PSQI score ≥6 (low perceived sleep quality)
* Medical questionnaire at baseline indicates they are healthy in the opinion of the Investigator
* Ability of the participant to comprehend the full nature and purpose of the study including possible risks and side effects in the opinion of the Investigator
* Agreement to comply with the protocol and study restrictions
* Available for all study visits
* Agreement to refrain from heavy drinking, late-night alcohol and late-night caffeine during the study
* Females of child-bearing potential required to provide a negative urine pregnancy test
* Easy access to internet, using email on a daily basis.

Exclusion Criteria:

* Any known history of a disorder affecting sleep quality, such as narcolepsy, obstructive sleep apnea (OSA), restless leg syndrome (RLS), periodic limb movement syndrome (PLMS) or any condition which contraindicates, in the Investigator's judgement, entry to the study
* Self-reported diagnosis of one or more DSM-V axis 1 disorder(s), including but not limited to current depression, anxiety disorder, bipolar spectrum disorder or schizophrenia
* Have a significant acute or chronic coexisting illness or any condition which contraindicates entry to the study in the opinion of the Investigator
* Previous (last 4 weeks prior to screening) or current intake of psychoactive medication (anxiolytics, sedatives, hypnotics, anti-psychotics, anti-depressants, anti-convulsants, centrally acting corticosteroids, opioid pain relievers)
* History of use (within 1 month of the first visit) or current intake (from day of screening onwards) of medication or dietary supplements/oriental herbs that could influence sleep patterns or that the Investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results (e.g. melatonin, omega-3 dietary supplements, non-steroidal anti-inflammatory drugs (NSAIDS), over-the-counter (OTC) sleep medication (not categorized as sedatives, hypnotics or anti-depressants), anti-coagulants, proton pump inhibitors, anti-histamines, pseudoephedrine, cortisone, beta-blockers)
* Self-declared illicit drug users (including cannabis and cocaine) for 3 months prior to screening and during the intervention period
* Heavy smoking (>10 cigarettes/day)
* High caffeine intake (> 10 cups /day) (or equivalent caffeine intake from other caffeinated drinks e.g., tea, energy drinks),
* Work schedule that causes irregular sleep pattern (e.g. night shift)
* History of travel to a different time zone within 1 month of the first visit or/and during the study participation
* Pregnant or lactating female, or pregnancy planned during intervention period
* Not fluent in German
* Contraindication or allergy (e.g. fish allergy) to any substance in the investigational product
* Participation in another study with any investigational product within 30 days of screening and during the intervention period
* Investigator believes that the participant may be uncooperative and/or noncompliant and should therefore not participate in the study.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of sleep quality | 18 weeks
  Measured with the Pittsburgh Sleep Quality Index (PSQI) at each visit

SECONDARY OUTCOMES:
Duration of sleep | 18 weeks
  Measured by a daily online diary over the total study
Evaluation of anxiety | 18 weeks
  Measured with a questionnaire at each visit
Evaluation of perceived stress | 18 weeks
  Measured with a questionnaire at each visit
Evaluation of depression, anxiety and stress | 18 weeks
  Measured with a questionnaire at each visit
Evaluation of quality of life | 18 weeks
  Measured with a questionnaire at each visit
Evaluation of systolic and diastolic blood pressure | 18 weeks
  Measured at each visit

OTHER OUTCOMES:
Evaluation of salivary cortisol | 18 weeks
  Measured the day and evening prior to each visit

CONTACTS AND LOCATIONS:
Overall Officials: Juliane Hellhammer, PhD, Principal Investigator — Daacro
Locations (1):
- daacro GmbH & Co. KG, Trier, Germany

REFERENCES:
- [Derived] Eckert F, Meyer N, Monzel E, Bouvret E, Chataigner M, Hellhammer J. Efficacy of a fish hydrolysate supplement on sleep quality: A randomized, double-blind, placebo-controlled, crossover clinical trial. Clin Nutr ESPEN. 2024 Apr;60:48-58. doi: 10.1016/j.clnesp.2024.01.002. Epub 2024 Jan 13. PMID 38479939